CLINICAL TRIAL: NCT07211828
Title: Pharmacodynamic Effects of Propofol and Alfentanil on EEG During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: EEG and Pain Monitor Data Under Anesthesia to Study Pharmacodynamic Effects of Opioids and Sedatives
Acronym: SED-ERCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chi Kwan Fung (Other)
Collaborators: National Yang Ming Chiao Tung University (Other); WeiGong Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Chi Kwan Fung, Attendant Physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH114-REC2-080
Record Dates: First submitted 2025-08-31; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Sedation and Analgesia; Cholangiopancreatography, Endoscopic Retrograde; Anesthesia, General
Keywords: sedation; phramacodynamics; opioid; ERCP
MeSH Terms: conditions — Agnosia | interventions — Alfentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation with high dose of alfentanil with the presence of propofol (Experimental): Adjust dose of alfentanil until reaching to the upper limit before adjusting dose of propofol. This aims to have a highest dose of alfentanil during anesthesia.
  Interventions: Drug: high dose of alfentanil
- Sedation with low dose of alfentanil with the presence of propofol (Active Comparator): Adjust dose of propofol to the upper limit before adjusting dose of alfentanil. This aims to have alfentanil less or equal to 10ng/mL during anesthesia.
  Interventions: Drug: low dose of alfentanil with propofol

INTERVENTIONS:
Drug: high dose of alfentanil — The initial dose is alfentanil cet 10ng/mL and propofol 1ug/mL. Dose of alfentanil will be increased by 10ng/mL each until PSI reach to 25-50. If alfentail has been adjusted to 50 but PSI is still too high, increase propofol cet by 0.5-1ug/mL till target PSI is reached. If propofol is adjusted to 0 but PSI is still too low, decrease alfetanil by 10ng/mL The range of dosage of alfentanil is 0-50ng/mL while propofol is 0-5ug/mL.
  Other Names: Alfenta; Alfentanil hydrochloride; Propofol (Diprivan)
  Arms: Sedation with high dose of alfentanil with the presence of propofol
Drug: low dose of alfentanil with propofol — Adjust dose of propofol to the upper limit before adjusting dose of alfentanil. Increase dose of propofol 0.5-1 ug/mL in order to have PSI valued 25-50. The initial dose of propofol is 1ug/mL, alfentanil 10 ng/mL. If propofol was adjusted to cet=5 ug/mL but PSI is still too high, increase alfentanil by 10 ng/mL instead. If alfentanil was adjusted to 0 but PSI is still too low, decrease propofol by 0.5-1 ug/mL instead . The range of dosage of propofol is 0-5 ug/mL while alfentanil is 0-50ng/mL.
  Other Names: Propofol (Diprivan); Alfenta; Alfentanil hydrochloride
  Arms: Sedation with low dose of alfentanil with the presence of propofol

SUMMARY:
Recording and analyzing electroencephalogram (EEG) and continuous pain monitor data under anesthesia in order to investigating the pharmacodynamic effects of opioids and sedatives.

DETAILED DESCRIPTION:
The Patient State Index (PSI) is the main instrument used for monitoring brain waves during anesthesia. By using conductive patches to detect frontal lobe brainwave patterns, PSI helps assess the patient's depth of anesthesia. The Analgesia Nociception Index (ANI) is a heart rate variability (HRV)-based indicator that evaluates the activity of the autonomic nervous system (sympathetic and parasympathetic), thereby reflecting the patient's pain or stress response. PSI and ANI are often used together in anesthetized patients to avoid drug overdose.

Since opioids and sedative drugs interact with each other, different doses of opioids and sedatives have varying effects on brain waves, PSI, and ANI. This interaction has recently become a focus in anesthesiology and critical care medicine.

The purpose of this study is to use target-controlled infusion (TCI) to continuously administer opioids and sedative drugs, and to observe changes in the Patient State Index (PSI), raw EEG, and ANI data during the anesthesia process, in order to identify the effects of opioids and sedatives on PSI, EEG, and ANI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who under go ERCP who require general anesthesia

Exclusion Criteria:

* ASA> or = 4 , vulnerable groups such as prisoners, patients with physical or mental disabilities and HIV carriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-03-16 (Estimated)

PRIMARY OUTCOMES:
EEG alpha power to beta power ratio | Baseline and periprocedural
EEG alpha ratio | baseline and periprocedural
EEG delta ratio | baseline and periprocedural
EEG beta ratio | baseline and periprocedural
Patient State Index (PSI) | baseline and periprocedural
  A processed electroencephalogram (EEG) parameter derived from frontal EEG signals. It is being measured continuously by a EEG monitor.

SECONDARY OUTCOMES:
Analgesia Nociception Index (ANI) | Baseline and periprocedural
  The Analgesia Nociception Index is measured by a continuous analgesia monitoring system . It is a numeric index (range from 0-100) indicating patients' nociception.
Blood pressure | baseline and periprocedural
Non-invasive cardiac output | during the whole sedation
  Cardiac output measured continuously by non-invasive monitoring (e.g., electrical cardiometry or equivalent device). The unit of measure is liters per minute (L/min)
Heart rate | baseline and periprocedural
Peripheral Capillary Oxygen Saturation (SpO₂) | baseline and periprocedural
  Continuous non-invasive measured by pulse oximetry,
Non-invasive cardiac index | baseline and periprocedural
  Cardiac index calculated as cardiac output normalized to body surface area, measured non-invasively. The unit of measure is liters per minute per square meter (L/min/m²)
Non-invasive Stroke Volume (SV) | baseline and periprocedural
  Stroke volume measured non-invasively, defined as the volume of blood ejected from the left ventricle per heartbeat.

OTHER OUTCOMES:
Frequency of Patient Movement Events | Periprocedural
  The total number of movement events (defined as gross body motion, limb withdrawal, or head movement) recorded during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chi Kwan Boris Fung, MD, Principal Investigator — Wei Gong Memorial Hospital